CLINICAL TRIAL: NCT06910319
Title: Six Minutes Walk Test in Children on Regular Hemodialysis at Assiut University Children Hospital
Brief Title: Six Minutes Walk Test in Children on Regular Hemodialysis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Caroline Fayez Abdelmalak, Doctor, Assiut University
Other Study IDs: 6 minutes walk test
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate exercise tolerance and the reproducibility of the six minute walk test in children and adolescents with ESRD on regular hemodialysis and to compare their functional exercise capacities with reference values for healthy children. To investigate predictors of poor 6MWT performance in children on regular HD

DETAILED DESCRIPTION:
The six-minute walk test (6MWT) is a submaximal test that assesses the functional exercise capacities of healthy subjects or those with a chronic disease, as well as the effects of interventions, such as pulmonary rehabilitation or drug therapies. It can predict prognosis, mortality and morbidity in adults and children with lung and/or heart diseases . A study with of children with stage V chronic kidney disease (CKD) has used the 6MWT to demonstrate decreased exercise tolerance , which appears to be caused by several factors, such as anemia, metabolic acidosis, electrolyte imbalance, osteopenia, growth deficiency, malnutrition, inactivity, uremic muscle dysfunction and associated comorbidities . The findings of this study suggest that the 6MWT could be used as a clinical tool to monitor functional exercise capacity in children with kidney disease. The 6MWT is a sub-maximum effort test that is more representative of daily life activities than other effort tests and has low cost and easy applicability . The distance walked in the 6MWT shows an association with VO2 peak, making it a viable and safe alternative for patients who cannot tolerate the ergometric test .

ELIGIBILITY:
Inclusion Criteria:

* Children with ESRD who on regular hemodialysis at Assiut University Children Hospital .

Exclusion Criteria:

* Any subject with underlying primary cardio-pulmonary disease or condition that interfere with the walk test as hemiplegia and cerebral palsy.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The patient observed the researcher performing the test and then was instructed to walk as far as possible for 6- min and maintain a normal walking pace. Patients are able to interrupt the test if necessary. At each minute of walking the researcher communicated clearly and calmly how many minutes remained until the end of the test. In the end, the walked distance will be measured. HR, %HRmax, SpO2, SBP, and DBP delta values are to be measured before and after participating test.
  During the test the researcher will monitor the patient for untoward signs and symptoms while using a stop watch to calculate time of the walked distance.If the patient stops before the 6 minutes are up and refuse to continue or the researcher decide that they should not continue, the researcher must wheel the chair over for the patient to sit on, discontinue the walk and note on the worksheet the distance , the time stopped and the reason for stopping prematurely.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the reproducibility of the six-minute walk test in children and adolescents with end stage renal disease on regular dialysis | One year from may 2025 to may 2026

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam Badawy Ali, Assistant professor of pediat, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe FT, Koch VH, Juliani RC, Cunha MT. Six-minute walk test in children and adolescents with renal diseases: tolerance, reproducibility and comparison with healthy subjects. Clinics (Sao Paulo). 2016 Jan;71(1):22-7. doi: 10.6061/clinics/2016(01)05. PMID 26872080
- [Background] Lipkin DP, Scriven AJ, Crake T, Poole-Wilson PA. Six minute walking test for assessing exercise capacity in chronic heart failure. Br Med J (Clin Res Ed). 1986 Mar 8;292(6521):653-5. doi: 10.1136/bmj.292.6521.653. PMID 3081210
- [Background] Gayda M, Temfemo A, Choquet D, Ahmaidi S. Cardiorespiratory requirements and reproducibility of the six-minute walk test in elderly patients with coronary artery disease. Arch Phys Med Rehabil. 2004 Sep;85(9):1538-43. doi: 10.1016/j.apmr.2003.11.037. PMID 15375831
- [Background] Painter P. Physical functioning in end-stage renal disease patients: update 2005. Hemodial Int. 2005 Jul;9(3):218-35. doi: 10.1111/j.1492-7535.2005.01136.x. PMID 16191072
- [Background] Bittner V, Weiner DH, Yusuf S, Rogers WJ, McIntyre KM, Bangdiwala SI, Kronenberg MW, Kostis JB, Kohn RM, Guillotte M, et al. Prediction of mortality and morbidity with a 6-minute walk test in patients with left ventricular dysfunction. SOLVD Investigators. JAMA. 1993 Oct 13;270(14):1702-7. PMID 8411500
- [Background] Savci S, Inal-Ince D, Arikan H, Guclu-Gunduz A, Cetisli-Korkmaz N, Armutlu K, Karabudak R. Six-minute walk distance as a measure of functional exercise capacity in multiple sclerosis. Disabil Rehabil. 2005 Nov 30;27(22):1365-71. doi: 10.1080/09638280500164479. PMID 16372431
- [Background] Du H, Newton PJ, Salamonson Y, Carrieri-Kohlman VL, Davidson PM. A review of the six-minute walk test: its implication as a self-administered assessment tool. Eur J Cardiovasc Nurs. 2009 Mar;8(1):2-8. doi: 10.1016/j.ejcnurse.2008.07.001. Epub 2008 Aug 9. PMID 18694656
- [Background] Painter P, Krasnoff J, Mathias R. Exercise capacity and physical fitness in pediatric dialysis and kidney transplant patients. Pediatr Nephrol. 2007 Jul;22(7):1030-9. doi: 10.1007/s00467-007-0458-6. Epub 2007 Mar 20. PMID 17372771
- [Background] Takken T, Engelbert R, van Bergen M, Groothoff J, Nauta J, van Hoeck K, Lilien M, Helders P. Six-minute walking test in children with ESRD: discrimination validity and construct validity. Pediatr Nephrol. 2009 Nov;24(11):2217-23. doi: 10.1007/s00467-009-1259-x. Epub 2009 Jul 25. PMID 19633871
- [Background] Pattaragarn A, Warady BA, Sabath RJ. Exercise capacity in pediatric patients with end-stage renal disease. Perit Dial Int. 2004 May-Jun;24(3):274-80. PMID 15185776
- [Background] Weaver DJ Jr, Kimball TR, Knilans T, Mays W, Knecht SK, Gerdes YM, Witt S, Glascock BJ, Kartal J, Khoury P, Mitsnefes MM. Decreased maximal aerobic capacity in pediatric chronic kidney disease. J Am Soc Nephrol. 2008 Mar;19(3):624-30. doi: 10.1681/ASN.2007070773. Epub 2008 Jan 9. PMID 18184856
- [Background] Sethna CB, Salerno AE, McBride MG, Shults J, Paridon SM, Sharma N, Meyers KE, Leonard MB. Cardiorespiratory fitness in pediatric renal transplant recipients. Transplantation. 2009 Aug 15;88(3):395-401. doi: 10.1097/TP.0b013e3181aed7d1. PMID 19667944
- [Background] Lammers AE, Hislop AA, Flynn Y, Haworth SG. The 6-minute walk test: normal values for children of 4-11 years of age. Arch Dis Child. 2008 Jun;93(6):464-8. doi: 10.1136/adc.2007.123653. Epub 2007 Aug 3. PMID 17675356
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Solway S, Brooks D, Lacasse Y, Thomas S. A qualitative systematic overview of the measurement properties of functional walk tests used in the cardiorespiratory domain. Chest. 2001 Jan;119(1):256-70. doi: 10.1378/chest.119.1.256. PMID 11157613